CLINICAL TRIAL: NCT05441215
Title: A PHASE I, MULTIPLE DOSE, OPEN-LABEL PHARMACOKINETIC STUDY OF NIRMATRELVIR/RITONAVIR IN HEALTHY LACTATING WOMEN
Brief Title: A Study to Learn About the Medicine (PF-07321332 or Nirmatrelvir/Ritonavir) in Healthy Lactating Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C4671039; 2022-001020-15 (EudraCT Number)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Healthy Participants
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2); Lactation; COVID-19; Breastfeeding; Protease Inhibitor
MeSH Terms: conditions — Breast Feeding; COVID-19 | interventions — nirmatrelvir; nirmatrelvir and ritonavir drug combination; Ritonavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nirmatrelvir/ritonavir (Experimental): nirmatrelvir/ritonavir will be given by mouth two times a day as a tablet
  Interventions: Drug: nirmatrelvir; Drug: ritonavir

INTERVENTIONS:
Drug: nirmatrelvir — nirmatrelvir/ritonavir
  Other Names: PF-07321332/ritonavir
Drug: ritonavir — nirmatrelvir/ritonavir
  Other Names: PF-07321332/ritonavir

SUMMARY:
The main purpose of this study is to measure the level of active ingredient of the study medicine (nirmatrelvir) that is secreted in human breast milk when it is given to healthy breastfeeding women. The study medicine consists of two medicines, nirmatrelvir and ritonavir. We are seeking female participants who are:

* Actively breast-feeding (lactating) at least 12 weeks postpartum;
* Age between 18 to 55 years and not currently pregnant;
* Have a Body Mass Index (BMI): 17.5 kg/m2; and a total body weight >50 kg (110 lb).

Participants will take the study medicine by mouth for a total of 3 times over 2 days (2 morning doses and 1 evening dose) at the study clinic. We will periodically collect breast milk from day 2 to 4 to measure the level of nirmatrelvir and ritonavir in it. A safety follow up call will be conducted around 28-35 days from the last dose to monitor any reactions participants may have to the study medicine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy lactating females who are actively breast-feeding or expressing breast milk, at least 12 weeks post-partum and not currently pregnant between 18 and 55 years old
* Body Mass Index (BMI): 17.5 kg/m2; and a total body weight >50 kg (110 lb)
* Infants of women enrolled in the study must be able to feed successfully from a bottle or other age-appropriate alternative feeding method prior to the start of the study and must be able to tolerate infant formula if the mother does not have a supply of stored breast milk sufficient to cover the duration of the study
* Participants must be willing to temporarily discontinue breast feeding their infants for a total of 4.5 days (108 hours)
* Participants must be willing to regularly pump breasts throughout the study and express milk according to a schedule designed to maintain lactation throughout the study period

Exclusion Criteria:

* Positive test result (RT-PCR) for SARS-CoV-2 infection at the time of screening or Day -1
* Evidence or history of clinically significant findings
* History of febrile illness or mastitis within 5 days prior to the first dose of study medication
* Participants who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed
* Abnormal vital signs such as blood pressure, 12-lead electrocardiogram
* History of alcohol abuse and/or illicit drug use, tobacco use in excess of 5 cigarettes/day or 2 chews/day
* Blood donation within 60 days

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy lactating women
Enrollment: 8 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Maximum Breastmilk Concentration (Cmax) of nirmatrelvir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Time to Reach Maximum Breastmilk Concentration (Tmax) of nirmatrelvir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Area under the breastmilk concentration time profile from time 0 to the time of the end of the dosing interval (tau) of nirmatrelvir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Terminal phase half life (t½) of nirmatrelvir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Average breastmilk concentration (Cav) of nirmatrelvir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Amount excreted in breast milk over the dosing interval (Aetau) of nirmatrelvir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Percent of dose excreted in breast milk during the dosing interval (Aetau %) of nirmatrelvir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Breast milk clearance (CLbm) of nirmatrelvir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)

SECONDARY OUTCOMES:
Cmax of ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Tmax of ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Area under the breastmilk concentration time profile from time 0 to the time of the end of the dosing interval (Auc tau) of ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
t½ of ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Cav of ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Aetau of ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Aetau % of ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
CLbm of ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Cmax of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Cav of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Pre-dose concentration (Ctrough) of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Tmax of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
AUC tau of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Minimum Observed Breastmilk Concentration (Cmin) of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
t½ of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Apparent plasma clearance (CL/F) of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Apparent volume of distribution (Vz/F) of nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Daily (24 hour) amount of nirmatrelvir excreted in breast milk (Ae 24bm) | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Breast milk to plasma ratio for AUC tau (MPAUC tau) for both nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Breast milk to plasma ratio for AUC tau (MPCmax during dosing interval tau) for both nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
CLbm for both nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Milk to plasma ratio (M/P) of both nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Body weight normalized infant dose in μg/kg/day (BWNID) of both nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Body weight normalized maternal dose in μg/kg/day (BWNMD) of both nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Infant dose expressed as % of body weight normalized maternal dose (BWNIDPCM) of both nirmatrelvir and ritonavir | Day 2 (0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours) and Day 3 (18, 24, 32, 40 hours) Day 4 (48 hours)
Participants reporting treatment emergent adverse events | Baseline to 28 days after last dose
Participants reporting abnormal clinical laboratory lab tests | Baseline to 28 days after last dose
Participants reporting abnormal vital signs | Baseline to 28 days after last dose
Participants reporting abnormal physical examination results | Baseline to 28 days after last dose
Participants reporting abnormal electrocardiograms | Baseline to 28 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671039